CLINICAL TRIAL: NCT00405054
Title: A Phase II Study of MK0457 in Patients With T315I Mutant Chronic Myelogenous Leukemia and Philadelphia Chromosome-positive Acute Lymphoblastic Leukemia
Brief Title: A Phase II Study of MK0457 in Patients With T315I Mutant CML and Ph+All (0457-008)
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0457-008; MK0457-008; 2006_551
Record Dates: First submitted 2006-11-28; First posted 2006-11-29 (Estimated); Last update posted 2015-01-26 (Estimated); Status verified 2015-01

CONDITIONS: Leukemia
MeSH Terms: conditions — Leukemia | interventions — tozasertib

ARMS (1):
- 1 (Other): continuous infusion every 14 days
  Interventions: Drug: MK0457

INTERVENTIONS:
Drug: MK0457 — IV infusion 32 mg/m2/hour; 5-day continuous infusion every 14 days

SUMMARY:
This study will evaluate MK0457 in patients with chronic myelogenous leukemia and Philadelphia chromosome-positive acute lymphoblastic leukemia. Efficacy and safety will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* This study will evaluate MK0457 in patients with CML (chronic myelogenous leukemia) and Ph+ALL (Philadelphia chromosome-positive acute lymphoblastic leukemia)
* Patients must have adequate organ function
* Patients must have documented T315I mutation

Exclusion Criteria:

* Patients within 3 months of allogeneic bone marrow transplant or not fully recovered from previous anti-leukemia therapy
* Patients with uncontrolled congestive heart failure
* Patients with active or uncontrolled infection or active Hepatitis B or C
* Patients with known HIV positivity or AIDS related illness
* Patients with currently active second malignancy, other than non-melanoma skin cancer.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2006-12; Primary Completion 2009-06 (Actual); Study Completion 2009-06 (Actual)

PRIMARY OUTCOMES:
efficacy | 24 Months

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC

REFERENCES:
- [Result] Seymour JF, Kim DW, Rubin E, Haregewoin A, Clark J, Watson P, Hughes T, Dufva I, Jimenez JL, Mahon FX, Rousselot P, Cortes J, Martinelli G, Papayannidis C, Nagler A, Giles FJ. A phase 2 study of MK-0457 in patients with BCR-ABL T315I mutant chronic myelogenous leukemia and philadelphia chromosome-positive acute lymphoblastic leukemia. Blood Cancer J. 2014 Aug 15;4(8):e238. doi: 10.1038/bcj.2014.60. PMID 25127392